CLINICAL TRIAL: NCT01916278
Title: A Randomized, Evaluator-blinded, Comparative Study of the Safety and Efficacy of Lip Injections With Emervel Lips Lidocaine and Juvéderm Volbella With Lidocaine
Brief Title: Safety and Efficacy Study of Lip Injections With Emervel Lips Lidocaine and Juvéderm Volbella With Lidocaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Other Study IDs: 05DF1215
Record Dates: First submitted 2013-07-18; First posted 2013-08-05 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2015-09

CONDITIONS: Lip Filler Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Emervel Lips Lidocaine (Experimental)
  Interventions: Device: Emervel Lips Lidocaine
- Juvéderm Volbella with Lidocaine (Experimental)
  Interventions: Device: Juvéderma Volbella with Lidocaine

INTERVENTIONS:
Device: Emervel Lips Lidocaine
  Arms: Emervel Lips Lidocaine
Device: Juvéderma Volbella with Lidocaine
  Arms: Juvéderm Volbella with Lidocaine

SUMMARY:
A 12-month, randomised, evaluator-blinded, comparative, multicentre study of the safety and efficacy of lip injections with Emervel Lips Lidocaine and Juvéderm Volbella with Lidocaine.

ELIGIBILITY:
Inclusion Criteria:

* Female and male subjects aged 18 to 65 years.
* Subjects with the intention to undergo lip augmentation treatment (vermilion mucosa and, if applicable, vermilion borders).
* Subjects with LFGS score of 0 (very thin), 1 (thin) and 2 (moderately thick) (scores may differ between upper and lower lip), and lip appearance judged by the treating investigator to be suitable for optimal correction (≥ 1 grade improvement on the LFGS per lip) with maximum 1.5 mL study product per lip.
* Subjects with signed informed consent.

Exclusion Criteria:

* Concomitant anticoagulant therapy and therapy with inhibitors of platelet aggregation (e.g. aspirin or other nonsteroidal anti-inflammatory drugs [NSAIDs]), Omega-3 or vitamin E within 10 days before study treatment, or a history of bleeding disorders.
* Prior surgery or tattoo to the upper or lower lip or lip line.
* Presence of any abnormal lip structure, such as a scar or lump or severe lip asymmetry, as judged by the investigator. Tendency to form keloids, hypertrophic scars or any other healing disorders.
* Previous tissue augmenting therapy in the lip area (including lips, oral commissures, nasolabial folds, marionette and perioral lines) with HA or collagen filler, or laser treatment, within 12 months before study entry.
* Permanent implant or treatment with non-HA or non-collagen filler in the lip area (including lips, oral commissures, nasolabial folds, marionette and perioral lines).
* Previous toxin treatment below the lower orbital rim within 9 months before study entry.
* History of herpes labialis with an outbreak within 4 weeks of study entry or with 4 or more outbreaks in the 12 months before study entry.
* Active skin disease, inflammation or related conditions, such as infection, psoriasis and herpes zoster near or on the area to be treated.
* History of angioedema.
* Known hypersensitivity to HA, lidocaine or other amide-type anaesthetics or history of severe multiple allergies or anaphylactic shock
* Cancerous or precancerous lesions in the area to be treated.
* Immunosuppressive therapy, chemotherapy, treatment with biologics or systemic corticosteroids within 3 months before study treatment.
* Any medical condition that in the opinion of the investigator would make the subject unsuitable for inclusion (e.g. a chronic, relapsing or hereditary disease that may affect the general condition or may require frequent medical treatment).
* Pregnancy or breast feeding.
* Participation in any other clinical study within 30 days before inclusion.
* Other condition preventing the subject to entering the study in the investigator's opinion, e.g. subjects not likely to avoid other facial cosmetic treatments below the level of the lower orbital rim and chin, subjects anticipated to be unreliable or incapable of understanding and complying with the study assessment or unrealistic expectations of treatment result.
* Study site staff or close relatives to study site staff and employees at the sponsor company or close relatives to employees at the sponsor company. Close relatives are defined as parents, children, siblings and spouse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2013-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Lip Fullness Grading Scale (LFGS) score | 0-12 months
  To evaluate esthetic change of lips from baseline using LFGS

OTHER OUTCOMES:
Global Aesthetic Improvement Scale (GAIS)score | 1-12 months
  To evaluate esthetic change of lips from baseline using GAIS
Subject's satisfaction | 0-12 months
  To evaluate subject's satisfaction in terms of a subject satisfaction questionnaire
Investigator's assessment of treatment procedure | 0-2 weeks
  To evaluate the ease of injection and moulding
Local tolerability | 14 days
  To assess local tolerability after treatment including bruising, redness, swelling, pain, tenderness and itching at 14 days. Local tolerability ongoing 2 weeks after treatment will be recorded as an AE and continued follow-up.
Subject's assessment of treatment pain | 0-2 weeks
  To evaluate subject's experience of pain during treatment.
Product palpability | 0-2 weeks
  To evaluate if study product is palpable or not palpable. If assessed as palpable, also to evaluate if the feel is expected/normal or unexpected/abnormal. Unexpected feel of palpable product present 2 weeks after treatment will be recorded as an AE and continued follow-up.
Adverse Event reporting | 0-12 months
  To evaluate long-term safety throughout the study period

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (2):
  - Rosenpark Research, Darmstadt
  - Medical Skin Center, Düsseldorf
- Akademikliniken, Stockholm, Sweden